CLINICAL TRIAL: NCT03262701
Title: Custom Tray Application of Peroxide Gel as an Adjunct to Scaling and Root Planing in the Treatment of Periodontitis: A 6-Month Randomized Trial
Brief Title: Adjunctive Hydrogen Peroxide for Periodontal Therapy
Acronym: AHP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5180025
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis, Chronic
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydrogen Peroxide gel for 13weeks (Experimental): Subjects will receive the standard of care which is conventional non-surgical therapy for chronic periodontitis and be given 1.7% hydrogen peroxide gel, oral, 0.75g, twice-daily for 15 minutes for 13 weeks.
  Interventions: Drug: Hydrogen Peroxide Gel, 13 weeks
- Hydrogen Peroxide gel for 26weeks (Experimental): Subjects will receive the standard of care which is conventional non-surgical therapy for chronic periodontitis and be given 1.7% hydrogen peroxide gel, oral, 0.75g, twice-daily for 15 minutes for 26 weeks.
  Interventions: Drug: Hydrogen Peroxide Gel, 26 weeks
- Scaling and Root Planing (Other): Subjects will receive the standard of care which is conventional non-surgical therapy for chronic periodontitis without any interventional hydrogen peroxide application in one or two visits.
  Interventions: Other: Scaling and Root planing group

INTERVENTIONS:
Drug: Hydrogen Peroxide Gel, 13 weeks — 13 weeks of twice-daily use of custom tray application of 1.7% peroxide gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis.
  Other Names: Perio Protect®; 1.7% hydrogen peroxide gel
  Arms: Hydrogen Peroxide gel for 13weeks
Drug: Hydrogen Peroxide Gel, 26 weeks — 26 weeks of twice-daily use of custom tray application of 1.7% peroxide gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis.
  Other Names: Perio Protect®; 1.7% hydrogen peroxide gel
  Arms: Hydrogen Peroxide gel for 26weeks
Other: Scaling and Root planing group — Subjects will receive the standard of care which is conventional non-surgical therapy for chronic periodontitis without custom tray application of 1.7% peroxide gel
  Other Names: SRP group control
  Arms: Scaling and Root Planing

SUMMARY:
There have been many adjunctive treatments for the additional clinical benefits to scaling and root planing (SRP) in the treatment of chronic periodontitis. Topical hydrogen peroxide (HP) delivered in a custom fabricated tray has been shown to improve pocket depth (PD) and inflammation. The purpose of this study is to assess the adjunctive treatment outcome of HP gel in custom tray application in individuals with chronic periodontitis receiving SRP. The purpose of this investigator-initiated study is to evaluate and compare the clinical effects of scaling and root planing (SRP) combined with local delivery of 1.7% hydrogen peroxide (HP) gel in customized trays to that of SRP alone.

DETAILED DESCRIPTION:
Hydrogen peroxide (HP) has been used in for wound debridement and oral rinses in dentistry for a few decades. It is widely available in a bottle of 3% in liquid. The use of hydrogen peroxide in gel type in 1.7% as an adjunct to conventional periodontal therapy has been introduced but there are limited information on the efficacy. The current study is to design to evaluate the adjunctive treatment outcome of hydrogen peroxide gel in custom tray application in individuals with chronic periodontitis receiving non surgical therapy, scaling and root planing(SRP). To test the adjunct effect of HP gel in tray, there will be three parallel arms, one with the gel for the period of 26 week, one with the gel for 13 weeks and control group without the gel.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who can read and sign the Research Information and Consent Form
2. Male and female adults, aged ≥18 years.
3. The presence of twenty or more (at least 2 posterior teeth in contact per quadrant, one of which is a molar), natural teeth in a good state of repair with scorable surfaces.
4. Show evidence of chronic periodontitis, minimum of one site with PD ≥5mm and Bleeding on Probing (BOP) in at least two quadrants and no mechanical debridement for six months prior to the start of the study.
5. Agree to comply with the conditions and schedule of the study, i.e., willing to use the assigned products (see Treatment Phase and Standardize Oral Hygiene Instruction) according to instructions and be available for appointments.
6. Agree not to have a dental prophylaxis, professional whitening treatment, or any other elective, non-emergency dental procedure (other than those provided) at any time during the study.
7. Willing to refrain from using mouth rinses and tooth whitening products for the duration of the study.

Exclusion Criteria:

1. Any systemic conditions or medication intake that can alter periodontal status (e.g. uncontrolled diabetes (with <3 month recent HbA1c of >8.5%), anti-seizure medication and immunosuppressants, and calcium channel blockers with clinical evidence of drug-influenced gingival enlargement)
2. Immune-compromised state.
3. Any current heavy smoking habits (>10 cigarettes/day)
4. Any medical condition or history requiring prophylactic antibiotic coverage prior to dental treatment.
5. Females who are lactating or pregnant (as determined by medical history) or planning to become pregnant for the duration of the study.
6. Physical limitations/restrictions compromising oral hygiene procedures.
7. The presence of significant oral soft tissue pathology and/or lesions associated with ill-fitting appliances or restorations.
8. Tooth mobility associated with advanced periodontal disease (e.g. score of >2 using Miller Classification).
9. Any temporomandibular joint disorders.
10. Grossly carious, orthodontically banded, and third molars will not be included in the tooth count.
11. The presence of any significantly tipped, crowded, or largely defective restorations.
12. Any extreme adverse events relating to the use of hydrogen peroxide gel (e.g. prolonged

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jeong Kim, DDS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Started | 14 | 17 | 9
Completed | 11 | 13 | 8
Not Completed | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing | Total
Number analyzed (Participants) | 14 | 17 | 8 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 6 | 33
  >=65 years | 1 | 3 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.5) | 54.5 (15.4) | 57.1 (15.7) | 52.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 4 | 19
  Male | 6 | 10 | 4 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 17 | 8 | 39
Bleeding On Probing [Mean (Standard Deviation); unit: percent] | 57.1 (37.2) | 66.9 (11.9) | 35.2 (16.8) | 53.1 (22.9)
Pocket Depth [Mean (Standard Deviation); unit: millimeters] | 4.11 (1.43) | 3.41 (1.16) | 3.82 (1.29) | 3.78 (1.29)
Relative Attachment Level [Mean (Standard Deviation); unit: millimeters] | 6.97 (1.29) | 7.11 (0.83) | 6.75 (0.16) | 6.94 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Periodontal Pocket Depth Reduction
Description: Periodontal pocket depth reduction as measured by the periodontal probe from the gingival margin to the bottom of the periodontal pocket measured in millimeters.
Time Frame: Change between baseline and Week 4
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Number analyzed (Participants) | 11 | 13 | 8
millimeters | -0.05 (0.16) | -0.16 (0.05) | 0.05 (0.09)

2. Primary Outcome: Periodontal Pocket Depth Reduction
Description: as for outcome 1
Time Frame: Change between baseline and Week 13
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Number analyzed (Participants) | 11 | 13 | 8
millimeters | -0.69 (0.31) | -0.54 (0.33) | -0.34 (0.09)

3. Primary Outcome: Periodontal Pocket Depth Reduction
Description: as for outcome 1
Time Frame: Change between baseline and Week 26
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Number analyzed (Participants) | 11 | 13 | 8
millimeters | -0.70 (0.33) | -0.49 (0.21) | -0.30 (0.14)

4. Secondary Outcome: Change in Clinical Attachment Level
Description: Change in clinical attachment level measured by using a periodontal probe with a stent used for reproducible reference in millimeters.
Time Frame: Change between baseline and Week 26
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Number analyzed (Participants) | 11 | 13 | 8
millimeters | -0.25 (0.65) | -0.42 (0.13) | -0.23 (0.16)

5. Secondary Outcome: Change in Bleeding on Probing
Description: Change in bleeding on probing measured by the presence of bleeding upon probing a periodontal pocket using a periodontal probe within 30 seconds measured in percentage.
Time Frame: Change between baseline and Week 26
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
Number analyzed (Participants) | 11 | 13 | 8
percent | -24.1 (23.2) | -34.2 (5.95) | -14.2 (10)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Hydrogen Peroxide Gel for 13weeks | Hydrogen Peroxide Gel for 26weeks | Scaling and Root Planing
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17 | 0/8
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17 | 0/8

LIMITATIONS AND CAVEATS:
Due to COVID lockdown, the enrollment and study discontinued abruptly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT03262701/Prot_SAP_000.pdf